CLINICAL TRIAL: NCT03040219
Title: Folic Acid Supplementation as an Appetizer in Primary Malnourished Egyptian Infants and Children
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Marian girgis, Principal investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 27111982
Record Dates: First submitted 2017-01-20; First posted 2017-02-02 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Primary Malnurtrition
MeSH Terms: interventions — Folic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Treatment group (Active Comparator)
  Interventions: Drug: Folic Acid
- Control (Placebo Comparator)
  Interventions: Drug: Folic Acid

INTERVENTIONS:
Drug: Folic Acid — Tablets

SUMMARY:
Folic acid as a appetizer in primary malnutrition

ELIGIBILITY:
Inclusion Criteria:

Primary malnourished children

Exclusion Criteria:

* previous folic supplementation in the past 3 months

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2017-04-01 (Estimated); Primary Completion 2017-11-01 (Estimated); Study Completion 2017-12-01 (Estimated)

PRIMARY OUTCOMES:
Appetite | Through study completion_ after 3 months from start of supplementation
  Child eating behaviour questionnaire

SECONDARY OUTCOMES:
Leptin and ghrelin hormone | 3 months
  Serum level

OTHER OUTCOMES:
Growth | Through study completion -after 3 months from start of supplementation
  Anthropometric study

CONTACTS AND LOCATIONS:
Overall Officials: Marian Girgis, Principal Investigator — Ain Shams University
Locations (1):
- Marian girgis, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided